CLINICAL TRIAL: NCT03832413
Title: Characterization of the DELPhI System in Assessing Brain's Functionality in Different Neurological Disorders-A Pilot Study
Brief Title: Characterization of the DELPhI System in Assessing Brain's Functionality in Different Neurological Disorders
Status: Completed | Type: Observational
Sponsor: QuantalX Neuroscience (Industry)
Responsible Party: Sponsor
Other Study IDs: QuantalX_pilot_asaf_harophe
Record Dates: First submitted 2018-11-01; First posted 2019-02-06 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2019-02

CONDITIONS: Stroke; TBI; Fibromyalgia; PDD; Adhd; ABD; Ptsd; Healthy; MCI; Dementia; Cognitive Impairment; Cognitive Decline
MeSH Terms: conditions — Stroke; Fibromyalgia; Attention Deficit Disorder with Hyperactivity; Stress Disorders, Post-Traumatic; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (10):
- Stroke: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- TBI: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- ABD: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- Fibromyalgia: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- PDD: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- ADHD: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- MCI: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- Dementia: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- Healthy: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)
- Cognitive impairment: Diagnostic Test: DELPhI (TMS-EEG analysis)
  Interventions: Diagnostic Test: DELPhI (TMS-EEG analysis)

INTERVENTIONS:
Diagnostic Test: DELPhI (TMS-EEG analysis) — We perform an evaluation not an intervention. the DELPhI evaluation comprises of an automated analysis to EEG data recorded during TMS (Transcranial Magnetic Stimulation) to the M1L (Primary motor cortex).

SUMMARY:
We use Transcranial magnetic stimulation (TMS), combined with simultaneous registration of electroencephalograph (EEG),for examining human cortical functionality. TMS-EEG is a noninvasive brain stimulation method that allows to study human cortical function in vivo. EEG provides an opportunity to directly measure the cerebral response to TMS, measuring the cortical TMS Evoked potential (TEP). In this study we measure TEPs, in a wide variety of neurological conditions and healthy as a measure of cerebral reactivity across wide areas of neocortex.

DETAILED DESCRIPTION:
Brain network plasticity evaluation has been shown extensively essential for understanding and monitoring of brain functional changes and brain disorders. However, existing clinically used imaging methods are unable to robustly indicate plasticity or plasticity changes. Therefore, there is a great need for developing such an imaging tool for brain functional evaluation. In basic neuroscience research plasticity evaluation is performed by conducting electrophysiological measurements in vivo. By using EEG - combined with TMS stimulation this methodology can be transformed into clinically used plasticity and connectivity assessment for evaluation of functional brain status. This study may thus introduce a novel, non-invasive and efficient method for brain functional imaging. DELPhI evaluation will offer a true multimodality imaging by combining EEG and TMS that allows a quantative objective and direct identification of disease assessment. There is a real unmet need for an accurate and objective evaluation that together with the common clinical practice will provide neurologists and psychiatrists a more definite and personalized treatment prescription.

Studies integrating TMS with EEG (TMS-EEG) have shown that TMS produces waves of activity that reverberate throughout the cortex and that are reproducible and reliable thus providing direct information about cortical excitability and connectivity with excellent time resolution. By evaluating the propagation of evoked activity in different behavioral states and in different tasks, TMS-EEG has been used to causally probe the dynamic effective connectivity of human brain networks. When applying the TMS coil above the motor cortex, a cascade effect called the motor-evoked potential (MEP), is initiated. The MEP is measurable at peripheral muscles. The Motor cortex is a brain structure located between the frontal and parietal cortices. Pyramidal neurons in the motor cortex, upper motor neuron going through the brain stem, send signals to lower motor neuron in the spinal cord which stimulate muscle fibers. TMS stimulus to the Motor cortex evokes a brain response which propagates to different brain regions in addition to the peripheral limb muscles [20]. An important feature of TEP topography is that even though only one cortical hemisphere is stimulated, bihemispheric EEG evoked responses are evoked with different features. TMS-evoked activity propagates from the stimulation site ipsilaterally via association fibers and contralaterally via transcallosal fibers and to subcortical structures via projection fibers. These TMS-evoked cortical potentials (TEPs) last for up to 300 ms in both the vicinity of the stimulation as well as in remote interconnected brain areas reflect long term changes in cortical network excitation-inhibition balance refeed to as brain network plasticity. A single TMS pulse delivered over the primary motor cortex (M1) results in a sequence of positive and negative EEG peaks at specific latencies (i.e., P25, N45, P70, N100, and P180).

In this study a wide population of subjects will be recruited. this population will include different neurological conditions and healthy subjects, arriving to the Hyperbaric center at Asaf-Harophe hospital. Each subject will be tested once before treatment initiation and subsequent tests will be performed also after treatment termination or at follow up time points. Each evaluation will last up to 90 minutes and will include affixed stimulation protocol ranging Up to 1000 TMS pulses, with intensities between 60-130% of motor threshold (MT). Inter-stimuli frequency will change from 0.01 up to 20 Hz.Existing clinical data such as MRI scans, neurocognitive assessments and clinical evaluations will be collected out of patient files. EEG data recorded will be analyzed and corrolations to the clinical data will be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Man and woman at the ages of ≥18 years.
2. Designated to perform a neurocognitive evaluation at the Sagol center for hyperbaric medicine and research, at Assaf-Harofe Medical center.

Exclusion Criteria:

1. Under 18 years of age.
2. With a skin condition on the scalp preventing the placement of EEG cap.
3. Pregnant or breastfeeding woman.
4. Unable to give an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients arriving to the Sagol center for Hyperbaric medicine at Assaf harofe Medical center, undergoing a series of hyperbaric treatment sessions and will be found compatible to inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Correlation between DELPhI's parameters to MRI scans | through study completion, an average of 1 year
  Correlation between DELPhI parameters to cognitive assessment by MRI/CT and computerized cognitive evaluation (Mindstreems cognitive battery test).
Correlation between DELPhI's parameters to cognitive assessment | through study completion, an average of 1 year
  Correlation between DELPhI parameters to MRI/CT and computerized cognitive evaluation (Mindstreems cognitive battery test).

SECONDARY OUTCOMES:
Cluster TMS Evoked Responses' (TEPs') features such as amplitude, latency, Area under the curve and slopes. | through study completion, an average of 1 year
  Calculating potential clusters based on TEP's features at different stimulation conditions. Features such as amplitude, area under the curve, slope and latency.

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf-Harophe, Rishon LeZiyyon, Israel